CLINICAL TRIAL: NCT03810833
Title: A Study of Tolerability and Background Fluorescence of the MediBeacon Transdermal GFR Measurement System
Brief Title: Tolerability and Background Fluorescence of the MediBeacon Transdermal GFR Measurement System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ORFM Sensor 100-01
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Acute Kidney Injury
Keywords: Glomerular Filtration Rate
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Participants with Brilliance sensor placement (Experimental): Brilliance device sensors placed on the left and right pectoralis major, remaining for 48 hours
  Interventions: Device: Brilliance device sensor

INTERVENTIONS:
Device: Brilliance device sensor — Two separate sensors will be attached via standard, single-use adhesive pads to the left and right pectoralis major on each participant.

SUMMARY:
This study is designed to evaluate background fluorescence of participants of different ages, gender, and skin color. In addition, 48-hour tolerability of the sensor and adhesive will be evaluated.

DETAILED DESCRIPTION:
The MediBeacon Transdermal GFR Measurement System investigational is intended to measure the Glomerular Filtration Rate (GFR) in patients with normal or impaired renal function by noninvasively monitoring fluorescent light emission from an exogenous tracer agent (MB-102) over time. The device utilized in this study is the Brilliance device. Approximately 1 male and 1 female from each age cohort (18-50 years; 51+ years) and clustered Fitzpatrick Skin Scale groups (I-II [Light, pale white; white, fair]; III-IV [Medium, white to olive; olive, moderate brown]; and V-VI [Brown, dark brown; black, very dark brown to black]) will be recruited, for a total of 12 participants. Participants will have Brilliance device sensors placed on two locations on their skin, which will remain for 48 hours. The sensor location will be prepared through shaving and cleaning (as applicable), placed on the skin via standard single-use adhesive pads, and baseline measurements collected. Participants may undergo activities of daily living while measurements are being collected. Light pressure and other minor perturbations may be applied to the sensors to evaluate the effect on background fluorescence. Adverse events associated with sensor placement (such as skin irritations) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults age 18 and older
* 2 age cohorts to be recruited: 18 - 50 years of age and 51+ years or older
* Skin color groups to be recruited in accordance with the Fitzpatrick Skin Scale (I - VI)
* Participants willing to sign the Institutional Review Board (IRB) approved informed consent form prior to the initiation of any study specific procedures.

Exclusion Criteria:

* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Significant scarring, tattoos or alterations in pigmentation on the standardized sensor locations that would alter sensor readings versus other areas of the skin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Mean Background Fluorescence | From the time of sensor placement to 48 hours after placement
  Two separate Brilliance device sensors will be attached via standard adhesive pads to the left and right pectoralis major on each participant. Fluorescence measurements will be collected directly by the MediBeacon Transdermal GFR Measurement System Brilliance device, and will be continuously collected throughout the 48 hour study.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon
Locations (1):
- St. Louis Clinical Trials, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No